CLINICAL TRIAL: NCT04011826
Title: The Evaluation of a New Nasal Mask for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-262
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Results first posted 2021-07-06 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: After a period of baseline, all enrolled participants will be put on the same trial mask.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental: Experimental trial nasal mask (Experimental): Experimental trial nasal mask: Participants will be placed on this arm for a total of 14±3 days from Visit 2. Participants will be using the trial nasal mask during this treatment arm. Participants on the extension will use this trial mask for a further six months after Visit 3.
  Interventions: Device: Device: Trial nasal mask (F&P)

INTERVENTIONS:
Device: Device: Trial nasal mask (F&P) — This trial nasal mask will serve as the participant's primary PAP/BPAP therapy mask for the duration of the trial period (from Visit 2 to Visit 3). For participants taking part in the study extension, they will be using the trial nasal mask as their primary PAP/BPAP therapy mask for 6 months after Visit 3.
  Other Names: New nasal mask

SUMMARY:
This investigation is designed to evaluate the comfort, ease of use and performance of a trial nasal mask for the treatment of Obstructive Sleep Apnea (OSA) in the home environment.

DETAILED DESCRIPTION:
The investigation is a prospective, non-randomized, non-blinded study. Up to 45 OSA participants who currently use a nasal, sub-nasal or pillows mask will be recruited.

The study will involve a baseline (Visit 1) data gathering with the participant's PAP therapy and their usual mask. This will be followed by the participants being fitted with the trial nasal mask by a mask fitting expert for use in-home (Visit 2). There will be a follow up phone call to gain feedback or address any issues after 3±1 days. The participant will then come in to return the mask (Visit 3) and give feedback on their experience using the mask in home in the form of a structured interview during Visit 3. If the participants prefer the trail nasal mask they will be asked if they would like to continue using the trial mask for a further six months in-home. There will be a follow up monthly phone call to gain feedback or address any issues during the extension. At the end of the six month extension period, the participants will return the trial nasal mask to the institution and give feedback on their experience using the mask in home in the form of a self-administered questionnaire. Participants will revert to their usual masks thereafter. Neither the participants nor the investigators will be blinded to the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OSA by Physician
* ≥ 22 years of age
* ≥ 66 lbs
* Prescribed PAP or BPAP therapy for OSA
* Existing nasal, sub-nasal and pillows mask users
* Fluent in written and spoken English

Exclusion Criteria:

* Inability to give informed consent
* Pregnant or think they may be pregnant
* PAP Intolerant
* Anatomical or Physiological Conditions that make PAP inappropriate
* IPAP pressure of ≤25cmH20.
* PAP/BPAP therapy device without data recording capabilities
* Using a PAP/BPAP therapy device for the delivery any medication with the exception of oxygen

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Muehlbach, Principal Investigator — Clinical Director
Locations (1):
- Clayton Sleep Institute, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with any other researchers or organizations.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: Experimental Trial Nasal Mask
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Experimental Trial Nasal Mask
Number analyzed (Participants) | 45
Age, Customized [Count of Participants; unit: Participants]
  Age 22+ years | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 32
  Other ethnicity (Hispanic/African American/Asian/Polynesian Descent | 13
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Objective Trial Mask Performance
Description: Objective measure (determined from efficacy data recorded from the participants PAP/BPAP therapy device.
  Adequate therapy was evaluated by reviewing the Apnea Hypopnea Index (AHI) at baseline to intervention within each individual participants from their PAP therapy device reports. Maintenance of therapy was determined by evaluating the change in AHI. The below data demonstrates how many participants of the analyzed population demonstrated maintenance of therapy after using the new F&P nasal mask.
Time Frame: 14 ± 3 days in home
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Experimental Trial Nasal Mask
Number analyzed (Participants) | 42
Participants | 42

2. Secondary Outcome: Number of Participants Trial Mask Overall Simplicity of Use
Description: Determined from questionnaires - Subjective (uses a 5-point Likert scale measuring ease of use, from very simple, simple, average, challenging, very challenging). Results below represent percentage of respondents for each value.
Time Frame: 14 ± 3 days in home
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Experimental Trial Nasal Mask
Number analyzed (Participants) | 45
percentage of participants
  Very Simple | 53
  Simple | 36
  Average | 2
  Challenging | 7
  Very Challenging | 2

3. Secondary Outcome: Number of Participants Subjective Trial Mask Comfort
Description: Determined from questionnaires - Subjective (uses a 5-point Likert scale measuring comfort from very comfortable, comfortable, average, uncomfortable, very uncomfortable). Participants reported their subject views on mask comfort. Responses to each likert scale option are presented below as percentages.
Time Frame: 14 ± 3 days in home
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Experimental Trial Nasal Mask
Number analyzed (Participants) | 45
percentage of participants
  Very comfortable | 39
  Comfortable | 37
  Average | 11
  Uncomfortable | 11
  Very uncomfortable | 2

4. Secondary Outcome: Number of Participants Overall Trial Mask Satisfaction
Description: Determined from questionnaires and a sleep diary - Subjective (measuring overall mask satisfaction, includes discussion, questions around overall satisfaction and preference of the new F&P Nasal mask compared to participants' usual mask ).
Time Frame: 14 ± 3 days in home
Population: A data size of 44 was used for this analysis due to missing data for one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Experimental Trial Nasal Mask
Number analyzed (Participants) | 44
Participants
  Preferred F&P nasal mask | 24
  Did not prefer F&P nasal mask | 20

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Experimental: Experimental Trial Nasal Mask
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 5/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Experimental Trial Nasal Mask (N=45)
Sinus Headaches (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rawness on side of nose (Skin and subcutaneous tissue disorders) | 1 (1)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain in Left Leg (General disorders) | 1 (1)
Pre-scheduled Cataract Surgery (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT04011826/Prot_001.pdf